CLINICAL TRIAL: NCT01948635
Title: Impact of Tracheal Cuff Shape on Microaspiration in Intensive Care Units
Acronym: BestCuff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012_45; 2013 A00534 41 (Other: ID-RCB number, ANSM); PHRCI_2012 (Other: PHRC numner, DGOS)
Record Dates: First submitted 2013-08-31; First posted 2013-09-23 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2018-05

CONDITIONS: Critical Illness; Mechanical Ventilation Complication; Ventilator Associated Pneumonia
Keywords: tracheal cuff shape; microaspiration; pepsin; ventilator-associated pneumonia
MeSH Terms: conditions — Critical Illness; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tapered PVC-cuffed tracheal tubes (Experimental): Patients in this arm will be intubated with tapered PVC-tracheal tubes
  Interventions: Device: tapered PVC-cuffed tracheal tubes
- Standard PVC-cuffed tracheal tube (Active Comparator): Patients in this arm will be intubated with standard (barrel-shape cuffed) PVC tracheal tubes
  Interventions: Device: Standard PVC-cuffed tracheal tube

INTERVENTIONS:
Device: tapered PVC-cuffed tracheal tubes — Patients will be intubated with tapered-shape tracheal tubes
  Arms: tapered PVC-cuffed tracheal tubes
Device: Standard PVC-cuffed tracheal tube — Patients will be intubated with standard PVC cuffed tracheal tubes
  Arms: Standard PVC-cuffed tracheal tube

SUMMARY:
The investigators hypothesized that PVC tapered-cuff tracheal tubes would reduce microaspiration of gastric content as determined by pepsin level in tracheal aspirate.

DETAILED DESCRIPTION:
Microaspiration is the main route for entry of contaminated secretions into the lower respiratory tract of intubated critically ill patients. Tracheobronchial colonization might progress to ventilator-associated pneumonia (VAP) when the quantity and virulence of bacteria are high and when local and general host defenses are weak.

Recent in vitro and animal studies suggest that tapered-cuff tracheal tubes could be associated with reduced microaspiration of contaminated secretions and might be helpful in preventing VAP.

ELIGIBILITY:
Inclusion Criteria:

* age > or = 18 years
* tracheal intubation
* predictable duration of mechanical ventilation > 48h
* enteral nutrition

Exclusion Criteria:

* pregnant women
* refuse to participate to the study
* no informed consent
* contre indication for semirecumbent position

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2014-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Microaspiration of gastric contents | 48 hours after randomization
  Mesuerment of pepsin level in tracheal aspirate will be used to quantify microaspiration of gastric contents

SECONDARY OUTCOMES:
Microaspiration of oropharyngeal secretions | 48 h after randomization
  amylase level on tracheal aspirate would allow to quantify microaspiration of oropharyngeal secretions
Tracheobronchial colonization | 28 days after randomization
Ventilator-associated pneumonia | 28 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Saad Nseir, MD, PhD, Principal Investigator — CHRU de Lille
Locations (9):
- France (9):
  - ICU, Salengro Hospital, University Hospital of Lille, Lille, Nord
  - centre Hospitalier, Boulogne-sur-Mer
  - Centre Hospitalier, Dunkirk
  - Centre Hospitalier, Lens
  - Centre Hospitalier St Philibert, Lomme
  - Centre hospitalier, Roubaix
  - Centre Hospitalier Universitaire, Rouen
  - Centre Hospitalie, Tourcoing
  - Centre Hospitalier, Valenciennes

REFERENCES:
- [Background] Jaillette E, Brunin G, Girault C, Zerimech F, Chiche A, Broucqsault-Dedrie C, Fayolle C, Minacori F, Alves I, Barrailler S, Robriquet L, Tamion F, Delaporte E, Thellier D, Delcourte C, Duhamel A, Nseir S. Impact of tracheal cuff shape on microaspiration of gastric contents in intubated critically ill patients: study protocol for a randomized controlled trial. Trials. 2015 Sep 25;16:429. doi: 10.1186/s13063-015-0955-z. PMID 26407612
- [Result] Jaillette E, Girault C, Brunin G, Zerimech F, Behal H, Chiche A, Broucqsault-Dedrie C, Fayolle C, Minacori F, Alves I, Barrailler S, Labreuche J, Robriquet L, Tamion F, Delaporte E, Thellier D, Delcourte C, Duhamel A, Nseir S; BestCuff Study Group and the BoReal Network. Impact of tapered-cuff tracheal tube on microaspiration of gastric contents in intubated critically ill patients: a multicenter cluster-randomized cross-over controlled trial. Intensive Care Med. 2017 Nov;43(11):1562-1571. doi: 10.1007/s00134-017-4736-x. Epub 2017 Mar 16. PMID 28303301